CLINICAL TRIAL: NCT05248347
Title: An Efficacy of Simulator Training for Fiberbronchoscopy in Intensivists
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Principal Investigator, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20220116ZDSYZYJ
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Simulator Training
Keywords: Fiberbronchoscopy; Simulation; Assessment; Validity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bronchoscopy training simulator (Active Comparator): Bronchoscopy training simulator LM-092 (Koken Co., Ltd, Tokyo, Japan) was used to train the participants.
  Interventions: Device: Bronchoscopy training simulator LM-092 (Koken Co., Ltd, Tokyo, Japan)
- The BRONCH Mentor (Experimental): Group B: The BRONCH Mentor (Simbionix, GI-Bronch Mentor, USA) was used.
  Interventions: Device: The BRONCH Mentor (Simbionix, GI-Bronch Mentor, USA)

INTERVENTIONS:
Device: Bronchoscopy training simulator LM-092 (Koken Co., Ltd, Tokyo, Japan) — Participants who passed the theory test and was enrolled in this group will use this device to practice. After the appropriate time of practice, the test will be taken to evaluate the efficacy.
  Arms: Bronchoscopy training simulator
Device: The BRONCH Mentor (Simbionix, GI-Bronch Mentor, USA) — Participants who passed the theory test and was enrolled in this group will use this device to practice. After the appropriate time of practice, the test will be taken to evaluate the efficacy.
  Arms: The BRONCH Mentor

SUMMARY:
We evaluated the effects of different fiberbronchoscopy training in how to teach and assess performance. Resident participants with no experience of fiberbronchoscopy, and doctors with little clinical experience with fiberbronchoscopy were eligible for the study.

DETAILED DESCRIPTION:
Participants who passed the theory test were enrolled in the study, and two training simulators for fiberbronchoscopy were used. After randomization, participants were enrolled in Group A (Bronchoscopy training simulator LM-092 )and Group B(The BRONCH Mentor). The test will be taken after practice at the appropriate time.

ELIGIBILITY:
Inclusion Criteria:

Doctors with little experience of fiberbronchoscopy

Exclusion Criteria:

* Resident participants who can not complete the study.
* Resident participants who can not pass the theroy examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Final score for examination by Bronchoscopy training simulator | through study completion, an average of 3 months
  Final score of manipulation, orientation, anatomy and actual operation

SECONDARY OUTCOMES:
% time at mid-lumen for fiberbronchoscopy manipulation by Bronchoscopy training simulator | through study completion, an average of 3 months
  % time at mid-lumen for fiberbronchoscopy manipulation by Bronchoscopy training simulator
% time at mid-lumen | through study completion, an average of 3 months
  % time at mid-lumen
% time at mid-lumen for fiberbronchoscopy manipulation | through study completion, an average of 3 months
  % time at mid-lumen for fiberbronchoscopy manipulation
Total wall hits for fiberbronchoscopy manipulation by Bronchoscopy training simulator | through study completion, an average of 3 months
  Total wall hits for fiberbronchoscopy manipulation by Bronchoscopy training simulator

CONTACTS AND LOCATIONS:
Overall Officials: Jingyuan Xu, M.D., Study Director — Southeast University
Locations (1):
- Nanjing Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided